CLINICAL TRIAL: NCT05757076
Title: Aldosterone Renin Ratio (ARR) Test to Increase Case-detection of Primary Aldosteronism (PA)
Acronym: ARR
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-132
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Screening Cohort: This is a prospective specimen collection cohort study aimed to increase the detection of primary aldosteronism (PA) in patients with hypertension.
  Study samples will be obtained longitudinally. One collection of plasma will be obtained. Blood draw may need to be repeated in some subjects after washout period. Study will continue for a period or 1 year, with plan to enroll around 50 subjects.
  Interventions: Procedure: Blood test for ARR

INTERVENTIONS:
Procedure: Blood test for ARR — Blood test for calculating aldosterone and renin ratio (ARR)

SUMMARY:
The mission of this project is to increase the detection of Primary Aldosteronism (PA), the most common cause of secondary hypertension, which can either be cured surgically or treated with targeted medications.

DETAILED DESCRIPTION:
The mission of this project is to increase the detection of Primary Aldosteronism (PA), the most common cause of secondary hypertension, which can either be cured surgically or treated with targeted medications. It is caused by the autonomous secretion of aldosterone by the adrenal glands.

Hypertension, elevated adrenal aldosterone secretion, and suppressed renin are the hallmarks of PA. The prevalence of PA varies approximately from 5% up to 20%.

Clinicians continue to erroneously learn that PA is a very rare disorder, thus PA continues to be under-recognized and undertreated. PA is a major public health issue, and the current case-detection rate is much below the prevalence rates reported in studies. Correctly identifying PA in patients will enable effective treatment and potential cure for this disease Hypertension by itself is a major driver of cardiovascular morbidity and mortality. There are ~ 1 billion people diagnosed with hypertension in the world, and even if we take a conservative prevalence of PA of 5% amongst this population, it would yield a staggering number of 50 million.

Cardiovascular and cerebrovascular morbidity and mortality rates are higher in those with PA compared to patients with blood pressure-matched essential hypertension.

As per the current Endocrine Society Guidelines, only patients who meet specific clinical profiles are considered to be candidates for screening for PA. Typically screening involves a blood test for calculating aldosterone and renin ratio (ARR). An abnormal test indicates the possibility of PA. It is estimated that only 1% of patients are detected by these screening guidelines.

Given the underdiagnosed state of this condition, and the high cardiovascular, cerebrovascular, and renal risks it entails, we should broaden the population to be screened for PA. All patients with hypertension who are on at least one anti-hypertensive medication should be screened for PA, especially given the benefits from specific surgical or medical treatment.

This would help reduce disease burden in a cost-effective manner and will impact the Care of Patients

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study
* Participants limited to subjects in the CCF
* Age between and inclusive of 18 and 65 years of age
* No gender exclusion
* Patients diagnosed with Essential Hypertension by ICD-10 code on at least two occasions in the previous six months, even if not on medications for hypertension
* Patients on a single anti-hypertensive medication for at least six months with the diagnosis of hypertension

Exclusion Criteria:

* Those on a mineralocorticoid antagonist therapy (spironolactone, eplerenone)
* Those with a documented diagnosis of primary aldosteronism or primary hyperaldosteronism
* Those with a diagnosis of secondary hyperaldosteronism
* Those with a diagnosis of heart failure, renal artery stenosis, cirrhosis, ascites, cor pulmonale.
* Pregnancy status (verbal)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled prospectively, under Institutional Review Board (IRB) approval and patient informed consent. Enrollment will include patients with known hypertension diagnosed via ICD-10 code who are on a single anti-hypertensive medication. Primary Care Physicians will identify potential patients and they will discuss with patients the possibility of participating in the study. The PCP will subsequently refer any potential patients that meet the criteria to the study team. A study coordinator will reach out to the patient via telephone encounter, MyChart message or mail to discuss the study in more detail. . Subjects will be consented in an office visit.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with Primary Aldosteronism (PA) that were missed. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No